CLINICAL TRIAL: NCT06505603
Title: Alpha-1 Antitrypsin PiMZ Longitudinal Cohort (PiMZ Logic)
Brief Title: PiMZ Longitudinal Cohort (PiMZ Logic)
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Alpha-1 Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: AAAU9605
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Alpha 1-Antitrypsin Deficiency; Emphysema or COPD
Keywords: Alpha-1; Biomarker; PiMZ
MeSH Terms: conditions — alpha 1-Antitrypsin Deficiency; Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Genetic sequencing and analysis may be performed on the DNA or RNA in some samples (blood and nasal swab). The biological samples may be prepared and, in some cases, analyzed at the Irving Institute for Clinical and Translational Research, the UCLA Nasal Swab Biorepository, or the Institute of Genomic Medicine of Columbia University. The purpose of the genetic testing is to find out any genetic (inherited) trait that would make participants more likely to have lung injury. A clause in the consent form addresses future use of data and specimens and participants have a choice to accept or decline this use.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Emphysema: FEV1/FVC <70%

SUMMARY:
Alpha-1 Anti-trypsin Deficiency (AATD) is a genetic disease with lung and liver disease presentations. Presentations are variable in the heterozygous population, the most predominant genotype being PiMZ. The purpose of this study in PiMZ heterozygous patients is to examine the density of the lung as measured by chest computed tomography (CT) and determine if existing emphysema predicts changes in the rate of subsequent emphysema or changes in CT, serum or plasma biomarkers of interest. The overarching goal is to develop biomarkers pertinent to the PiMZ patient that can be used in interventional trials since lung function changes do not typically inform disease progression in AATD.

DETAILED DESCRIPTION:
Progression of lung disease in patients with Alpha-1 Anti-trypsin deficiency is variable and while some patients may have stable lung function over many years, some progress and deteriorate rapidly. Currently there are no predictors that would help identify patient at risk of rapid deterioration in the PiMZ patient population. The aim of this study is to identify markers and features in CT imaging that may allow identification of these patients early before deterioration. To achieve this, the study will follow a cohort of patients with confirmed Alpha-1 Anti-trypsin deficiency (MZ genotype) and obstructive lung disease and measure a number of biomarkers in blood and sputum and obtain high resolution CT scans at baseline and again three years later. If the study is able to determine markers that allow the identification of patients at risk early, the investigator may be able to study early interventions in later studies and possibly find ways to avoid serious complications. Patients will be followed longitudinally to assess deterioration of lung function.

Study procedures include: Review of medical history and medication history, blood draw, spriometry, induced sputum (at some sites), completion of questionnaires and CT Chest scan. All of the mentioned procedures above will be performed on enrollment and repeated at 18 months and 36 months, with the exception of monthly Alpha- net exacerbation questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged 18 years and older
2. Understand the study procedures, risks, benefits, purpose
3. Able and willing to comply with the study procedures
4. Have PiMZ alpha-1 antitrypsin deficiency
5. Post bronchodilator FEV1 < 80% predicted AND post bronchodilator FEV1/FVC < 70%
6. Be an existing member of the Alpha-1 Foundation Clinical Cohort (also known as the Alpha-1 Foundation Research Registry)
7. Agree to have the data collected in this study be shared with the Alpha-1 Foundation Research Registry

Exclusion Criteria:

1. AATD non-PiMZ status, including carriers
2. Current lung, hematologic, or solid organ malignancy other than skin or cervical Stage 1 cancers within the past 3 years
3. COPD exacerbation or other pulmonary infection within 6 weeks of baseline visit
4. Pregnancy at the time of the screening visit
5. Inability to lie still in a supine position for 15 minutes during CT acquisition
6. Inability to perform quality-controlled lung function testing
7. Allergy to albuterol
8. Currently receiving intravenous or subcutaneous immunoglobulin for any disease state
9. Past or present major surgery on the lungs including pneumonectomy or lobectomy. Wedge resections, past segmentectomy, and pleurodesis surgeries are allowed.
10. Previous lung or liver transplantation or currently on the transplant list
11. Decompensated cirrhosis
12. Current presence of endobronchial coils or valves in the lung
13. Clinically significant bronchiectasis as defined by the investigator. In general, this would exclude patients with chronic infection of the lungs requiring treatment within the past 6 months including non-tuberculous mycobacterial disease, chronic fungal disease, allergic bronchopulmonary aspergillosis, or known colonization of bronchiectasis with pseudomonas or stenotrophomonas species.
14. Participation in the active treatment arm of a therapeutic clinical trial at baseline visit unless using one of the Alpha-1 augmentation therapies in alternative doses.
15. Patient with Automatic Implantable Cardioverter Defibrillator (AICD) and permanent pacemakers (PPM)
16. Patient receiving biologic immunomodulators that will affect the assessment of the serum biomarkers (as determined by the site PI)
17. Patient with pleural catheters
18. Any condition that in the opinion of the investigator might adversely influence the study outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Alpha-1 Antitrypsin Deficiency genotype MZ across the United States.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in lung density over three years | 3 years
  Change in lung density over three years determined by using the 15th percentile point (PERC-15) of Hounsfield units in inspiratory high resolution CT scans.
Decline of PERC-15 (15th percentile) over three years | 3 years
  Rate of decline of PERC-15 over three years. PERC-15 provides the Hounsfield unit point below which 15% of all voxels are distributed. The lowest threshold is -1,000 HU. The lower the PERC-15 values are, the more CT-quantified emphysema is present.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Goldklang, MD, Principal Investigator — Columbia University
Locations (5):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California- Los Angeles, Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - University of Chicago, Chicago, Illinois
  - Columbia University Irving Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: Yes
This study is part of a larger research study where one of the objectives is to create a AATD de-identified, public use repository of data. This repository will be query based, and any sub-projects that stem from this will need to abide by the appropriate Human Subjects Protection, GCP guidelines (i.e., IRB protocol, local IRB approval, DUA, Release of Information) and be reviewed by the research committee including the Alpha-1 Foundation prior to release of any de-identified data.
Supporting Information: Study Protocol
Time Frame: After first 3 years of data collection and preliminary analysis
Access Criteria: De-identified data will be available via i2b2 with proper protocol and IRB regulatory documentation.